CLINICAL TRIAL: NCT02697838
Title: Clinical Trial of Apatinib Reverses Chemotherapy-Resistance of Patients With Advanced Gastric Cancer
Status: Unknown | Phase: Phase 2 | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: Fujian Cancer Hospital (Other Government)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: AHEAD-G323
Record Dates: First submitted 2016-02-25; First posted 2016-03-03 (Estimated); Last update posted 2018-10-17 (Actual); Status verified 2018-10

CONDITIONS: Malignant Neoplasm of Stomach Stage II
MeSH Terms: conditions — Stomach Neoplasms | interventions — apatinib

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Experimental: Apatinib plus chemotherapy (Experimental)
  Interventions: Drug: Apatinib; Drug: Paclitaxel-based chemotherapeutic regimens

INTERVENTIONS:
Drug: Apatinib — Apatinib (850 mg qd p.o.) until disease progression or intolerable toxicity or refused by the patients.
Drug: Paclitaxel-based chemotherapeutic regimens — Paclitaxel-based chemotherapeutic regimens including:
  1. The POF regimen consisted of a 3-hour infusion of paclitaxel (135 mg/m2) followed by oxaliplatin (85 mg/m2) and Calcium Levofolinate (200 mg/m2).Subsequently, a 46-hour infusion of fluorouracil (2400 mg/m2) was administered using an ambulatory pump, repeating the cycle every 14 days.
  2. The PF regimen consisted of a 3-hour infusion of paclitaxel (135 mg/m2) followed by Calcium Levofolinate (200 mg/m2).Subsequently, a 46-hour infusion of fluorouracil (2400 mg/m2) was administered using an ambulatory pump, repeating the cycle every 14 days.
  3. Paclitaxel 80mg/m2 d1，d8，d15，repeating the cycle every 28 days
  4. other paclitaxel-based regimens

SUMMARY:
A single arm study: Apatinib plus paclitaxel as the reverses treatment in advanced gastric cancer which paclitaxel-resistant.

DETAILED DESCRIPTION:
This trial investigated the efficacy and safety of apatinib plus paclitaxel, as a treatment option for patients with advanced gastric cancer which paclitaxel-resistant.

ELIGIBILITY:
Inclusion Criteria:

1. Age: more than 18 years old;
2. Histologically confirmed advanced or metastatic adenocarcinoma of gastric cancer(AGC) , including adenocarcinoma of the gastroesophageal junction;
3. At least one measurable and evaluable disease based on response evaluation criteria in solid tumors (RECIST v1.1);
4. The patient with Prior Paclitaxel-Resistant;
5. Eastern Cooperative Oncology Group Performance Status (ECOG PS) of 0-2;
6. An expected survival of ≥ 3 months;
7. Duration from the last therapy is more than 6 weeks for nitroso or mitomycin, More than 4 weeks for other cytotoxic agents, operation or radiotherapy;
8. Major organ function has to meet the following criteria; (1) For results of blood routine test:

   1. Hemoglobin (HB) ≥ 80g / L,
   2. ANC ≥ 1.5 × 109 / L,
   3. PLT ≥ 75 × 109 / L, (2) For results of biochemical tests:

   <!-- -->

   1. BLT ≤ 1.25 times the upper limit of normal (ULN),
   2. ALT and AST ≤ 2.5 × ULN, liver metastases, if any, the ALT and AST≤ 5 × ULN,
   3. Serum Cr≤1ULN, Endogenous creatinine clearance rate >50ml/min;
9. Pregnancy test (serum or urine) has to be performed for woman of childbearing age within 7 days before enrolment and the test result must be negative. They shall take appropriate methods for contraception during the study until the 8th week post the last administration of study drug. For men, (previous surgical sterilization accepted), shall agree to take appropriate methods of contraception during the study until the 8th week post the last administration of study drug;
10. Patient has to voluntarily join the study and sign the Informed Consent Form for the study.

Exclusion Criteria:

1. History of other malignancies except cured basal cell carcinoma of skin and carcinoma insitu of uterine cervix;
2. Confirmed that apatinib and/or its accessories allergy;
3. Subjects with poor-controlled arterial hypertension (systolic blood pressure> 140 mmHg and diastolic blood pressure > 90 mm Hg) despite standard medical management;
4. Serious cardiovascular disease: Ⅱ-level myocardial ischemia or myocardial infarction, arrhythmia (including QT interval prolongation, for man ≥ 450 ms, for woman ≥ 470 ms); III ~ IV level cardiac function insufficiency, or echocardiography showed that left ventricular ejection fraction (LVEF < 50%);
5. Patients with positive urinary protein (urine protein detection of 2 or more, or 24 hour urine protein >1.0g);
6. Factors that could have an effect on oral medication (such as inability to swallow, chronic diarrhea and intestinal obstruction);
7. Subjects with high gastrointestinal bleeding risk, including the following conditions: local active ulcer lesions with positive fecal occult blood test (++); history of black stool, or vomiting blood in the past 2 months;unresected primary lesion in stomach with positive fecal occult blood test (+), ulcerated gastric carcinoma with massive alimentary tract bleeding risk judged by PIs based on gastric endoscopy result;
8. Abnormal Coagulation (INR>1.5、APTT>1.5 UNL), with tendency of bleed;
9. With psychotropic drug abuse history and can't get rid or with mental disorder patients;
10. Less than 4 weeks from the last clinical trial;
11. According to the researcher's judgment, with other serious diseases which harm to patient safety or affect patients complete the study;
12. Evidence of central nervous system(CNS) metastasis;
13. Pregnant or lactating women;
14. Other conditions regimented at investigators' discretion.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 20 (Actual)
Dates: Start 2016-08-01 (Actual); Primary Completion 2018-03-31 (Actual); Study Completion 2018-10-31 (Estimated)

PRIMARY OUTCOMES:
disease control rate(DCR) | 6 months

CONTACTS AND LOCATIONS:
Locations (1):
- Rongbo Lin, Fuzhou, Fujian, China

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Derived] Zhao S, Fan N, Li H, Liu J, Huang F, Chen Y, Zhou M, Yu J, Lin R. Apatinib combined with paclitaxel-based chemotherapy in patients with taxane-resistant advanced gastric cancer: a single-arm exploratory study. Ann Transl Med. 2020 Oct;8(19):1233. doi: 10.21037/atm-20-5841. PMID 33178765